CLINICAL TRIAL: NCT06912659
Title: Non-interventional Prospective Study in Patients With Pulmonary Fibrosis Treated With Nintedanib Participating in a Patient Support Program in Spain, to Describe Patient Satisfaction With the Program and to Monitor Quality of Life - BALANCE Study
Brief Title: The BALANCE Study: A Study in Spain to Find Out Whether a Patient Support Program Helps People With Pulmonary Fibrosis Who Take Nintedanib
Status: Active, not recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0575
Record Dates: First submitted 2025-04-03; First posted 2025-04-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients participating in the PSP Balance Program

SUMMARY:
The aim of this study is to describe patients' satisfaction with Patient Support Program (Balance Program), Quality of Life and depression symptoms, dosing pattern, disease symptoms, adverse events and nintedanib discontinuation (both permanent and non-permanent) from study inclusion to 12 months of follow-up.

ELIGIBILITY:
Inclusion criteria

* Adults (≥18 years old at baseline).
* Patients included in the Patient Support Program (PSP) Balance Program.
* Ability to read and speak Spanish correctly according to the investigator criteria.
* Agree to participate and signing informed consent at baseline.

Exclusion criteria

- Suspicion or diagnosis of any relevant cognitive impairment at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients with IPF and PPF (other than IPF) participating in the PSP Balance Program. The study duration will be from the start of the recruitment period (which will last approximately 6 months) to the last follow-up visit of the last patient (approximately 18 months of total study period). Patients will be followed-up at 6 months and at 12 months.
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with Patient Support Program (PSP) Balance Program at baseline using the Baker Questionnaire. | at Baseline
  Baker Questionnaire: This questionnaire contains 18 items divided into four domains. related to general satisfaction, the care provided by the professional, the time dedicated to the consultation and the relationship with the professional. There is no cut point published.
  Items in both modules have a five-option numeric score that ranges from 1 "Not at all" to 5 "Extremely". Total Baker score ranges from 0 to 90, with higher numbers indicating a greater satisfaction. In this study the mean value will be include.

SECONDARY OUTCOMES:
1. Change in the satisfaction with Patient Support Program (PSP) Balance Program at 6 and 12-month follow-up after inclusion in the study, using the Baker Questionnaire. | up to 12 months
  Baker Questionnaire: This questionnaire contains 18 items divided into four domains. related to general satisfaction, the care provided by the professional, the time dedicated to the consultation and the relationship with the professional. There is no cut point published.
  Items in both modules have a five-option numeric score that ranges from 1 "Not at all" to 5 "Extremely". Total Baker score ranges from 0 to 90, with higher numbers indicating a greater satisfaction. In this study the mean value will be include.
Patient satisfaction with PSP Balance Program at baseline, 6 and 12 months after the inclusion in the study using the Likert scale. | at baseline and up to 12 months
  Likert scale: This questionnaire contains 8 items. related to satisfaction with PSP, the care provided by the professional, the time dedicated to the consultation and the relationship with the professional. There is no cut point published.
  Items have a four-option numeric score that ranges from 1 "Not at all" to 4 "Extremely".
Dosing pattern of nintedanib calculated as absolute number of doses taken correctly divided by all the doses prescribed in that period (6 and 12 months) | up to 12 months
Time from first dose to permanent discontinuation of nintedanib within 12-month follow-up. | up to 12 months
Absolute number of nintedanib dose interruptions. | up to 12 months
Health-Related Quality of Life (HRQoL) at baseline and 12-month follow-up using the L-PF Impacts Questionnaire. | at baseline and up to 12 months
  Total score (from 0 to 100 points) and symptoms, impacts, dyspnea, cough and fatigue scores obtained in the L-PF Questionnaire at each visit
  L-PF Impacts Questionnaire:
  This questionnaire contains 44 items divided into two modules. The Impacts module (21 items) assesses multiple aspects of the quality of life with a recall period of 1 week. The questionnaire was developed recently (before it was used in Idiopathic Pulmonary Fibrosis (IPF) patients only) and there is no cut point published. The Symptoms module yields three domain scores: 1) dyspnea, 2) cough and 3) fatigue as well as a total Symptoms score. Items in both modules (L-PF Impacts and L-PF Symptoms) have a five-option numeric score that ranges from 0 "Not at all" to 4 "Extremely". Total L-PF score ranges from 0 to 100, with higher numbers indicating a greater impairment.
Anxiety and depression scores in Hospital Anxiety and Depression Scale (HADS) Questionnaire at baseline and 12-month follow-up. | at baseline and up to 12 months
  Total score (from 0 to 100 points) obtained in the HADS Questionnaire at each visit.
  HADS Questionnaire:
  The Hospital Anxiety and Depression Scale-Spanish Version is a 14-item self-report screening scale for anxiety and depression in Spanish-speaking populations. HADS consists of a 7-item anxiety subscale and a 7-item depression subscale. Each item scores on a 4-point Likert scale.
  Each item is scored on a scale of 0 = best to 3 = worst, which means that the maximum score for each subscale is 21. To interpret the results, the total sums of each subscale are considered separately. A score of 0 to 7 on any of the subscales is generally considered to be an absence of relevant disorder, 8 to 10 indicates the presence of borderline or borderline symptoms, and a score of 11 or higher suggests a significant presence of anxiety or depression.
Disease symptoms score in Living with Pulmonary Fibrosis (L-PF) Symptoms Questionnaire at baseline and 12 months follow-up. | at baseline and up to 12 months
  Total score (from 0 to 100 points) obtained in the L-PF Questionnaire at each visit.
  L-PF Symptoms Questionnaire:
  This questionnaire contains 44 items divided into two modules. The Symptoms module (23 items) rates shortness of breath, cough, and fatigue in the past 24 hours. The questionnaire was developed recently (before it was used in IPF patients only) and there is no cut point published.
  Items in both modules (L-PF Impacts and L-PF Symptoms) have a five-option numeric score that ranges from 0 "Not at all" to 4 "Extremely". Total L-PF score ranges from 0 to 100, with higher numbers indicating a greater impairment.
Absolute number of visits to emergency service and hospitalization related to Interstitial Lung Disease (ILD) between baseline and 12-month follow-up. | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Evidenze Health Espana S.L., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com